CLINICAL TRIAL: NCT05907837
Title: Early Detection & Intervention of Cerebral Palsy in Ireland
Status: Recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: National Maternity Hospital, Ireland (Other); University Maternity Hospital Limerick (Unknown); Cork University Maternity Hospital (Other); Coombe Women and Infants University Hospital (Other); The Rotunda Hospital (Other); Cerebral Palsy Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: EDI-CPI
Record Dates: First submitted 2023-06-02; First posted 2023-06-18 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Palsy; Neurodevelopmental Disorders
MeSH Terms: conditions — Cerebral Palsy; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (CP) is the most common lifelong physical disability. It is defined as a non-progressive disorder of movement originating from neural lesions in the perinatal period, and is associated with a wide range of common comorbidities in many individuals. These include problems speaking, hearing, seeing, thinking, feeding and controlling their bladder. People with CP often have additional challenges such as behavioural and emotional issues, pain, and poor sleep. Many of these challenges respond well to intervention in early childhood, as brain plasticity is at its greatest in the first 2 years of life. However, in most clinical settings, the age for diagnosis of CP is between 24 to 29 months, after this window of neurodevelopmental opportunity.

This project will aim to improve the Early Detection of Cerebral Palsy in Ireland. This will be achieved by implementing an evidence-based approach to follow-up of High risk infants.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardians must be able and willing to give written informed consent and to comply with the requirements of this study protocol.
* All infants considered high risk for cerebral palsy and neuro-developmental impairment will be eligible, specifically including:

  * All preterm infants born ≤32 weeks Post Menstrual Age or ≤1500 gm birth weight
  * All encephalopathic infants
  * Neurological risk factors (e.g., injury/malformation on neuroimaging, persistently abnormal neurological exam)

Exclusion Criteria:

* Death prior to discharge from the neonatal unit.

Max Age: 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns at high risk of developing CP will be identified and consented for inclusion prior to discharge from the Neonatal unit. Approximately 1500 infants will be recruited nationally over the study period from Cork University Maternity Hospital, University Maternity Hospital Limerick, The Coombe Hospital, The Rotunda Hospital and the National Maternity Hospital.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduce the age of CP diagnosis in Ireland. | 5 years
  Reduce the age of diagnosis of cerebral palsy in Ireland to less than 12 months of age by using evidence based standardised motor and neurological assessments at set time points.
Standardised Approach to Assessing infant at risk of CP | 5 years
  To establish a standardised approach to assessing infants at risk of CP in High Risk Follow-up Clinics across Ireland.

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Walsh, Principal Investigator — University College Cork; Breda Hayes, Principal Investigator — The Rotunda Hospital; Deirdre Sweetman, Principal Investigator — National Maternity Hospital; Roy Philips, Principal Investigator — Limerick University Maternity Hospital; John Kelleher, Principal Investigator — Coombe Women and Infants University Hospital
Locations (5):
- Ireland (5):
  - Cork University Maternity Hospital, Cork
  - Coombe Women and Infants University Hospital, Dublin
  - National Maternity Hospital, Dublin
  - The Rotunda Hospital, Dublin
  - University Maternity Hospital Limerick, Limerick

IPD SHARING:
Plan to Share IPD: No